CLINICAL TRIAL: NCT01421732
Title: Laboratory Diagnosis and Prognosis of Severe Dengue
Status: Completed | Type: Observational
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other); Children's Hospital Number 1, Ho Chi Minh City, Vietnam (Other); Number 2 Children's Hospital, Ho Chi Minh City (Other); Tien Giang Provincial Hospital, Tien Giang, Viet Nam (Unknown); Red Cross Clinic Of District 8 (Other)
Responsible Party: Sponsor
Other Study IDs: 13DX
Record Dates: First submitted 2011-08-22; First posted 2011-08-23 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Dengue Fever
Keywords: Dengue fever; severe dengue fever; NS1 detection assay; Prognosis; Diagnosis
MeSH Terms: conditions — Dengue; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected dengue fever: Children aged 1-15 presenting at participating hospitals with symptoms of dengue fever

SUMMARY:
A study of dengue in children presenting to outpatient departments of 5 large hospitals in Ho Chi Minh City and Tien Giang province, Viet Nam.

Different blood tests are compared at the early stages of dengue fever onset in their ability to accurately and specifically detect children whose dengue will progress to severe disease.

DETAILED DESCRIPTION:
In a prospective study in the outpatients department of three large hospitals in Ho Chi Minh City, Viet Nam, we will determine the early diagnostic sensitivity, specificity, positive and negative predictive values of two NS1 diagnostic tests in severe dengue cases.

The study is intended to develop a prognostic algorithm for the early identification of severe dengue cases.

Routine demographic, haematological and biochemical laboratory markers will be utilized to derive a prognostic algorithm that is clinically-useful for guiding patient triage and interventions.

We hope to discover and evaluate new early biomarkers of severe dengue and will evaluate candidate host response molecules and virological markers for their prognostic value.

We further plan to understand the phylogeography of DENV in the super-urban setting of HCMC.

We will use genome scale sequencing of DENV together with geospatial information on the residential addresses of patients to better understand transmission dynamics in space and time in a high transmission super-urban district of HCMC and thereby identify opportunities for public health interventions.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of dengue
* Axillary temperature >=37.5C
* Less than 72hrs of fever
* Resident in Ho Chi Minh City
* 1-15 yrs of age
* Accompanying family member or guardian has a mobile phone
* Written informed consent

Exclusion Criteria:

* Any patient who the attending physician believes is unlikely to be able to attend follow-up
* Any patient in who the attending physician believes another diagnosis is more likely.

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patient presenting to outpatient department of participating hospitals with symptoms of dengue fever
Sampling Method: Probability Sample
Enrollment: 8100 (Actual)
Dates: Start 2010-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the NS1 detection assays for diagnosis of laboratory-confirmed severe dengue. | Within the first 72 hours of fever onset
  Percentage of detection assays which correctly predict laboratory-confirmed severe dengue.
Specificity of the NS1 detection assays for diagnosis of laboratory-confirmed severe dengue. | Within the first 72 hours of fever onset
  Percentage of detection assays which correctly predict different dengue serotypes.
Positive predictive values of the NS1 detection assays for diagnosis of laboratory-confirmed severe dengue. | Within the first 72 hours of fever onset
  Percentage of detection assays which correctly predict dengue infection.
Negative predictive values of the NS1 detection assays for diagnosis of laboratory-confirmed severe dengue. | Within the first 72 hours of fever onset
  Percentage of detection assays which correctly predict no dengue infection.

SECONDARY OUTCOMES:
Positive predictive values of the NS1 detection assays for children requiring hospitalization or parenteral fluid therapy. | Estimated within 6 days of presentation
  Percentage of detection assays which correctly predict requirement of hospitalization and/or parenteral fluid therapy (dehydration, vomiting or signs of capillary permeability).
Negative predictive values of the NS1 detection assays for children requiring hospitalization or parenteral fluid therapy. | Estimated within 6 days of presentation
  Percentage of detection assays which correctly predict no requirement of hospitalization and/or parenteral fluid therapy (dehydration, vomiting or signs of capillary permeability).
Sensitivity of the NS1 detection assays to predict the requirement of hospitalization or parenteral fluid therapy. | Estimated within 6 days of presentation
  Percentage of detection assays which correctly predict the requirement of hospitalization and/or parenteral fluid therapy (dehydration, vomiting or signs of capillary permeability).
Specificity of the NS1 detection assays to predict the dengue serotype which corresponds to the requirement of hospitalization or parenteral fluid therapy. | Estimated within 6 days of presentation
  Percentage of detection assays which correctly predict the dengue serotype and it's correlation to a requirement of hospitalization and/or parenteral fluid therapy (dehydration, vomiting or signs of capillary permeability).

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Simmons, PhD, Principal Investigator — Oxford University Clinical Research Unit
Locations (1):
- Hospital for Tropical Diseases, Ho Chi Minh City, Ho Chi Minh, Vietnam

REFERENCES:
- See also: Oxford University Clinical Research Unit — http://www.oucru.org
- See also: Study details and Informed Consent Form — http://www.oucru.org/index.php?option=com_content&view=article&id=336&Itemid=111&lang=en